CLINICAL TRIAL: NCT03211637
Title: Implementing and Assessing an Wounds Protocol at Family Health Strategy Units in a Rio Grande do Sul Countryside Town
Brief Title: Wounds Protocol at Family Health Strategy Units in a Rio Grande do Sul Countryside Town
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Daniel Demétrio Faustino da Silva, PhD, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HNSConceicaoMP
Record Dates: First submitted 2017-02-27; First posted 2017-07-07 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Chronic Vascular Wounds in Adults
Keywords: nursing care; skin lesions; wound healing; varicose ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP (Experimental): This group comprises 6 healthcare units equipped with a Family Health Strategy, where patients are seen by coordinating nurses who have been trained to use wound dressing supplies and also on the use of the protocol.
  Interventions: Combination Product: Wounds Protocol
- CONTROL GROUP (Active Comparator): This group comprising 5 healthcare units equipped with a Family Health Strategy. Patients were seen by coordinating nurses who used techniques and supplies with which they were already familiar. They had no protocol in place.
  Interventions: Combination Product: Wounds Protocol

INTERVENTIONS:
Combination Product: Wounds Protocol — Nurses who have been trained to use wound dressing supplies and also on the use of the protocol.

SUMMARY:
Evaluate the process for implementing a wound protocol for lesion control and cost-effectiveness in the context of the Family Health Strategy in the city of Santa Cruz do Sul, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Presenting vascular (venous, arterial or mixed) ulcers for over 1 year;
* Be available to have wounds dressed at the healthcare unit;
* Be a patient registered with the Family Health Strategy teams.

Exclusion Criteria:

* Have some condition rendering the patient unable to go to the unit, such as being bedridden or having had a lower limb amputated;
* Having decompensated diabetes mellitus;
* Having move away from the Family Health Strategy unit's coverage area.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Lesion remission by measuring the surface area of the wound | one month
  Remission of the wound, and other clinical variables such as odor, pain, infection and presence of exudate.

IPD SHARING:
Plan to Share IPD: No